CLINICAL TRIAL: NCT00899873
Title: Proposed Study of CLL Samples
Brief Title: Biomarkers in Samples From Patients With Chronic Lymphocytic Leukemia Treated on Clinical Trial ECOG-2997
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000617494; ECOG-E2997T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cytogenetic Analysis; Flow Cytometry; Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: cytogenetic analysis
Other: flow cytometry
Other: fluorescence activated cell sorting
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of cells in the laboratory from patients with cancer may help identify biomarkers related to cancer. It may also help doctors learn how patients respond to treatment.

PURPOSE: This laboratory study is analyzing samples of cells from patients with chronic lymphocytic leukemia who were treated on clinical trial ECOG-2997.

DETAILED DESCRIPTION:
OBJECTIVES:

* To analyze the expression of a variety of informative molecules using a unique high-resolution flow cytometric immunophenotyping technology in samples from patients with chronic lymphocytic leukemia enrolled in clinical trial ECOG-2997.

OUTLINE: Cell samples are analyzed for the following prognostic biomarkers: ZAP-70, phospho-Syk, phospho-GSK-3β, phospho-Akt, phospho-ZAP-70, cyclin D1, cyclin D2, p21cip1, phospho-ReIA, IkappaBα, Bax, Mcl-1, PTEN, phospho-Erk1/2, and phospho-MEK1/2. Biomarker signals are amplified using enzymatic amplification staining to obtain high resolution detection of cell-surface markers on leukemic cells. Biomarker expression levels are measured using fluorescence activated cell sorting analysis. Relationships between clinical outcomes, standard flow cytometric analysis, cytogenetic studies, and high resolution immunophenotyping will also be assessed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Stored frozen viable cells from patients with chronic lymphocytic leukemia treated on clinical trial ECOG-2997

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients enrolled on E2997
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2012-04-17 (Actual); Primary Completion 2012-07-17 (Actual); Study Completion 2012-07-17 (Actual)

PRIMARY OUTCOMES:
Correlation of biomarker analysis and correlation with outcome response | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: David Kaplan, MD, PhD, Study Chair — University Hospitals Seidman Cancer Center